CLINICAL TRIAL: NCT00221702
Title: Randomized, Multicenter Phase III Trial Comparing Adjuvant Treatment With PegIntron Over 36 Months Versus Reference Treatment With IntronA Over 18 Months in Cutaneous Melanoma Patients AJCC Stage II (>=1.5 mm Clinically Node Negative)
Brief Title: PegIntron Versus IntronA in CMAJCC Stage II (EADO 2001/CMII Trial)
Acronym: EADO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Jean Pierre LEROY/ Clinical Research and innovation Director, University Hospital Bordeaux
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9267-01; 2001-034
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Melanoma; Neoplasm Metastasis
Keywords: Melanoma; Neoplasm metastasis; Interferon alfa-2b; Adjuvants; Randomized clinical trial; Disease-free survival time; Safety; Drug toxicity; Quality of life
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Drug-Related Side Effects and Adverse Reactions | interventions — peginterferon alfa-2b; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Peg Intron 100 mcg SC/week for 36 months
  Interventions: Drug: PegIntron
- B (Active Comparator): Intron A 3 X 3 MIU, weekly, sc, for 18 months
  Interventions: Drug: intron A

INTERVENTIONS:
Drug: PegIntron — 100 mcg SC/week for 36 months
  Arms: A
Drug: intron A — 3mui TIWW SC for 18 months
  Arms: B

SUMMARY:
Melanoma with a tumor thickness >= 1.5mm without clinically detectable nodes represents an increasing population with relapse rate of more than 50%. Adjuvant therapy with low doses of IFN alpha can provide a benefit in this group. However, the impact of low dose IFN alpha is not sustained after the treatment period. A longer treatment may prolong the benefit and thus have a more clear-cut impact on disease-free and overall survival. The tolerance and the impact on quality of life are limiting factors in a group of patients whose individual course is not necessarily poor. PegIntron may be better tolerated than instant release interferon, and thus make this treatment more acceptable in terms of toxicity and quality of life. Thus treatment schedule with PegIntron is not expected to increase the cost of standard care significantly.

DETAILED DESCRIPTION:
Study design and primary objective

This is an European multicenter, open label, prospective randomized phase III trial evaluating the efficacy of long-term maintenance therapy of two therapy options, IntronA for 18 months versus PegIntron for 36 months, administered in an adjuvant setting after the local excision of an intermediate risk cutaneous melanoma.

Eligibility criteria

Intermediate risk melanoma is defined by the following criteria: (1) a tumor thickness >= 1,5mm and (2) the absence of regional nodal macrometastases, as assessed either by clinical examination or, if sentinel lymph node biopsy (SLNB) or elective node dissection (ELND) are performed, by the absence of macroscopic evidence of disease. Patients with evidence of nodal micrometastasis by SLNB or ELND are eligible. The choice of performing sentinel node dissection will be left to the decision of each center, on condition to concern all consecutive patients and that all surgical procedures are completed before randomization of the patients . The centers have to inform their respective national study center if they perform SLNB or ELND and also if they change their surgical procedure.

Study treatments

* Arm A : PegIntron 100 mcg SC/week for 36 months
* Arm B : IntronA 3miu TIWW SC for 18 months

Endpoints

The primary endpoint of the study will be the time to any recurrence (local recurrence, satellite or in transit metastasis, regional node metastasis or distant metastasis) or death, whatever the cause. The primary comparison between the two arms will use the 5-year disease-free survival time. Secondary endpoints are time to distant metastasis , overall survival, toxicity and quality of life.

Therapy with either PegIntron or IntronA will continue as scheduled unless there is evidence of disease progression (whether local or distant recurrence), severe toxicity, or the subject requests that therapy be discontinued. All patients will be followed for disease-free-survival and overall survival until the end of the trial.

Sample size and analysis

The calculated sample size is 1190 patients to be enrolled over a 5 years period; this sample size is inclusive of an expected lost to follow up not more than 10% during the course of the trial. The randomization procedure will be stratified according to centers and to sentinel node biopsy. The primary analysis will be performed under the intent to treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cutaneous melanoma
* Tumour thickness >= 1.5 mm (Breslow staging)
* Absence of clinically detectable regional node metastasis, no evidence of distant metastasis
* Informed consent form signed

Exclusion Criteria:

* Any prior chemo-, immuno-, hormonal or radiation therapy
* Macroscopic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 898 (Actual)
Dates: Start 2003-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
disease-free survival time | 5-year

SECONDARY OUTCOMES:
time to distant metastasis | the time from the inclusion to the first documentation of any distant metastasis
overall survival | the time from the inclusion to the date of death regardless of the specific cause
toxicity | for 36 months
quality of life | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean - Jacques GROB, Professor, Principal Investigator — University Hospital, Marseille; Geneviève Chêne, Professor, Study Chair — University Hospital, Bordeaux
Locations (1):
- APHM, dermatology, Marseille, France

REFERENCES:
- [Derived] Grob JJ, Jouary T, Dreno B, Asselineau J, Gutzmer R, Hauschild A, Leccia MT, Landthaler M, Garbe C, Sassolas B, Herbst RA, Guillot B, Chene G, Pehamberger H. Adjuvant therapy with pegylated interferon alfa-2b (36 months) versus low-dose interferon alfa-2b (18 months) in melanoma patients without macrometastatic nodes: an open-label, randomised, phase 3 European Association for Dermato-Oncology (EADO) study. Eur J Cancer. 2013 Jan;49(1):166-74. doi: 10.1016/j.ejca.2012.07.018. Epub 2012 Sep 10. PMID 22975216